CLINICAL TRIAL: NCT04075734
Title: Promoting Follow-Up Care Self-Management for Adolescent and Young Adult (AYA) Childhood Cancer Survivors
Brief Title: Feasibility of a Self-Management + Peer Mentoring Intervention for Adolescent and Young Adult Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katie Devine, PhD, MPH, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20150001955; R21CA222936 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Childhood Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of (1) online self-management educational modules and (2) weekly peer mentor calls to facilitate engagement with the modules and offer specialized support over approximately six weeks.
  Interventions: Behavioral: Managing Your Health: Self-Management + Peer Mentoring
- Usual Care (No Intervention): Participants are not receiving the tested intervention. They continue to receive standard or routine psychosocial or transition care available to them as part of the normal practice

INTERVENTIONS:
Behavioral: Managing Your Health: Self-Management + Peer Mentoring — The online educational component consists of 5 self-management educational modules:
  (1) Understanding Your Survivorship Care Plan; (2) Managing Your Healthcare; (3) Family and Significant Other Involvement in Your Healthcare; (4) Emotions about Your Health and Follow-Up Care; (5) Staying Healthy.
  Participants will be matched with a peer mentor and complete a total of six calls. The first call is to build a rapport and identify the participant's self-management strengths, weaknesses, and goals. The next five calls align with the topic of each module, which the mentee is expected to complete prior to their scheduled call.
  Arms: Intervention

SUMMARY:
The goal of this project is to evaluate the feasibility of the "Managing Your Health" online self-management skills+peer mentoring intervention that focuses on overcoming survivor barriers to self-management of their survivorship care. We will conduct a pilot randomized controlled trial (RCT) of the intervention versus usual care with adolescent and young adult survivors of childhood cancer ages 18-25 years. Participants will complete survey measures at baseline, Time 2 (about 2 months after baseline), Time 3 (about 5 months after baseline), and Time 4 (about 12 months after baseline).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of the online self-management+peer mentoring program in a pilot RCT.

II. Assess preliminary efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Young Adult Survivors:

* age 18-25;
* at least 2 years from treatment for any pediatric cancer diagnosed at age 0-19;
* low self-reported responsibility for healthcare as indicated by reporting parent is primarily responsible for healthcare or low score (1 or 2) on two or more items from Readiness for Transition Questionnaire - Survivor Version.

Peer Mentor:

* age 21-29;
* at least 2 years from treatment for any pediatric cancer diagnosed at age 0-19;
* self-reported primary responsibility for healthcare and "complete" readiness to assume responsibility or high scores (3 or 4) on all items from Readiness for Transition Questionnaire - Survivor Version.

Exclusion Criteria:

• Documented or self-reported cognitive delay to prevent self-management of healthcare.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Devine, PhD, Principal Investigator — Rutgers Cancer Inst. of NJ
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The intervention consists of (1) online self-management educational modules and (2) weekly peer mentor calls to facilitate engagement with the modules and offer specialized support over approximately six weeks.
  Managing Your Health: Self-Management + Peer Mentoring: The online educational component consists of 5 self-management educational modules:
  (1) Understanding Your Survivorship Care Plan; (2) Managing Your Healthcare; (3) Family and Significant Other Involvement in Your Healthcare; (4) Emotions about Your Health and Follow-Up Care; (5) Staying Healthy.
  Participants will be matched with a peer mentor and complete a total of six calls. The first call is to build a rapport and identify the participant's self-management strengths, weaknesses, and goals. The next five calls align with the topic of each module, which the mentee is expected to complete prior to their scheduled call.
- Usual Care: Participants are not receiving the tested intervention. They continue to receive standard or routine psycho-social or transition care available to them as part of the normal practice.
- Mentors: Peer Mentors were recruited and matched 1:1 with each participant randomized to Intervention to facilitate engagement with the online modules and offer specialized support.
Period: Overall Study
Arm/Group | Intervention | Usual Care | Mentors
Started | 25 | 25 | 10
Completed | 21 | 24 | 10
Not Completed | 4 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RCT Intervention: The intervention consists of (1) online self-management educational modules and (2) weekly peer mentor calls to facilitate engagement with the modules and offer specialized support over approximately six weeks.
  Managing Your Health: Self-Management + Peer Mentoring: The online educational component consists of 5 self-management educational modules:
  (1) Understanding Your Survivorship Care Plan; (2) Managing Your Healthcare; (3) Family and Significant Other Involvement in Your Healthcare; (4) Emotions about Your Health and Follow-Up Care; (5) Staying Healthy.
  Participants will be matched with a peer mentor and complete a total of six calls. The first call is to build a rapport and identify the participant's self-management strengths, weaknesses, and goals. The next five calls align with the topic of each module, which the mentee is expected to complete prior to their scheduled call.
- RCT Usual Care: Participants receive usual care.
- Mentors: Peer Mentors were recruited and matched 1:1 with each participant randomized to RCT Intervention to facilitate engagement with the online modules and offer specialized support.
- Total: Total of all reporting groups
Arm/Group | RCT Intervention | RCT Usual Care | Mentors | Total
Number analyzed (Participants) | 25 | 25 | 10 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 10 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.12 (2.03) | 21.60 (1.89) | 26.50 (2.46) | 23.07 (2.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 5 | 25
  Male | 14 | 16 | 5 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 0 | 5
  Not Hispanic or Latino | 21 | 24 | 10 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 0 | 8
  White | 16 | 14 | 9 | 39
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 10 | 60

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Measure: Enrollment (Young Adult Survivors) - Number of Eligible Patients Consented and Completing Baseline
Description: Determined by number of eligible patients consented and completing baseline. Hypothesis: >50% of eligible will consent and complete the baseline.
Time Frame: Baseline
Population: All potentially eligible participants identified by the New Jersey State Cancer Registry (NJSCR) and approached at the local Long-Term Information Treatment Evaluation (LITE) program by study staff.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Control Trial Participants-Young Adult Survivors: Participants for the randomized trial (i.e., Young Adult survivors) were recruited using the New Jersey State Cancer Registry (NJSCR) and the local Long-Term Information Treatment Evaluation (LITE) program.
Arm/Group | Randomized Control Trial Participants-Young Adult Survivors
Number analyzed (Participants) | 79
Participants
  Enrolled | 50
  Not Interested | 29

2. Primary Outcome: Feasibility Measure: Retention in Study (Young Adult Survivors): Percent of Consented Patients Who Are Retained in the Study and Complete Time 3 Follow-up
Description: Retention in study (Young Adult Survivors). Determined by the percent of consented patients who are retained in the study and complete Time 3 follow-up. Hypothesis: >80%.
Time Frame: Time 3 at about 5 months since Baseline.
Population: Young Adult Survivors who enrolled on study, i.e., consented and completed baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
Participants | 22 | 25

3. Primary Outcome: Feasibility: Completion of the Intervention (Young Adult Survivors): Percentage
Description: Mean percent completed per task: (a) On-line self-management educational modules and (b) Weekly calls with peer mentor.
Time Frame: Time 2, about 2 months since baseline.
Population: Data available and reported only for participants who were assigned to this group and completed the tested intervention, i.e., n=22. Total of three participants assigned to this group, withdrew from the study, without completing the tested intervention.
Measure: Mean (Full Range); unit: percent completed
Arm/Group | Intervention
Number analyzed (Participants) | 22
percent completed
  On-line self-management educational modules | 95.72 [58.8 to 100]
  Weekly calls with peer mentor | 97.72 [66.7 to 100]

4. Primary Outcome: Feasibility: Satisfaction With Intervention (Young Adult Survivors): Mean
Description: Five items assess satisfaction with each aspect of the intervention: a. Overall program satisfaction; b. Content of online modules; c. Discussions with peer mentor; d. Frequency of calls with peer mentor; and e. Duration of program. First 3 items (a, b and c) were evaluated using a 5-point scale, (Minimum 1, Maximum 5) with higher scores indicating greater satisfaction. Item c evaluated on a scale from 1 "not frequent enough" to 3 "too frequent". Item d uses a 1 "way too short" to 5 "way too long" scale. The sample mean will be examined.
Time Frame: Time 2, about 2 months since baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 22
score on a scale
  a. Satisfaction w/ Program overall [Scale 1-5] | 4.64 (0.49)
  b. Satisfaction w/ Content of online modules [Scale 1-5] | 4.41 (0.59)
  c. Satisfaction w/ Discussions with peer mentor [Scale 1-5] | 4.64 (0.49)
  d. Satisfaction w/ Frequency of calls with peer mentor [Scale 1-3; 2="Just right"] | 2.00 (0.31)
  e. Satisfaction w/ Duration of program [Scale 1-5; 3= "Just right" | 2.86 (0.47)

5. Primary Outcome: Feasibility: Utility of the Online Self-Management Modules (Young Adult Survivors): Questionnaire
Description: The Utility Questionnaire is an 11-item scale that measures perceived ease of use and convenience of the online program using a 5-point scale, (minimum 1, maximum 5) with higher scores indicating greater perceived utility. An overall mean of all items will be calculated.
Time Frame: Time 2, about 2 months since baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 22
score on a scale | 4.35 (0.54)

6. Primary Outcome: Feasibility: Impact of the Online Self-Management Modules (Young Adult Survivors): Questionnaire
Description: The Impact Questionnaire is a 13-item scale that measures perceived effectiveness of the online program using a 5-point scale, (minimum 1, and maximum 5) with higher scores indicating greater perceived effectiveness. An overall mean of all items will be calculated.
Time Frame: Time 2, about 2 months since baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 22
score on a scale | 4.29 (0.48)

7. Primary Outcome: Feasibility: Adherence Barriers to the Online Self-Management Modules (Young Adult Survivors): Questionnaire
Description: The Adherence Barriers Questionnaire is a 6-item scale that measures perceived barriers to using the online program using a 5-point scale, (minimum 1 and maximum 5) with higher scores indicating greater perceived barriers. An overall mean of all items will be calculated.
Time Frame: Time 2, about 2 months since baseline.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 22
score on a scale | 1.17 (0.24)

8. Primary Outcome: Acceptance of Peer Mentors (Young Adult Survivors and Peer Mentors): Questionnaire
Description: Acceptance will be evaluated by young adult survivors' and peer mentors' report on perceived alliance with each other using the Working Alliance Inventory - Short Form Revised (Hatcher & Gillaspy, 2006), a validated measure of the quality and strength of the relationship. Items are rated on a 5-point scale. The measure yields 3 subscales summary scores that can range from 5 to 20, with higher scores indicating more positive relationships. Sum scores on each sub-scale with be calculated: Bond, Goal, and Task.
Time Frame: Time 2, about 2 months since baseline
Population: Peer mentors and young adult survivors in RCT Intervention group who completed the tested intervention (i.e., n=22). Please note, while total number of mentors on study was n=10, total reports by mentors for this measure was n=22 (some mentors were assigned to mentor more than one young adult survivor assigned to RCT intervention group.)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Mentors
Number analyzed (Participants) | 22 | 10
score on a scale
  Bond | 18.41 (1.92) | 19.55 (1.14)
  Goal | 17.68 (2.28) | 13.45 (1.71)
  Task | 18.14 (2.01) | 13.09 (1.66)

9. Secondary Outcome: Healthcare Responsibility (Young Adult Survivors)
Description: The Readiness for Transition Questionnaire - Survivor Version (RTQ) assesses the degree to which survivors are responsible for 10 healthcare behaviors, including knowing their survivorship care plan, scheduling annual visits, scheduling specialist appointments, taking and filling medications (if prescribed), explaining medical history to others, knowing insurance coverage, attending appointments, communicating with providers, and calling providers, on a 4-point scale, with higher scores indicating higher levels of responsibility. The RTQ yields a total mean score for responsibility. It also has one item evaluating "overall readiness to assume complete responsibility for healthcare" with response options of Not at all ready, somewhat ready, mostly ready, or completely ready. The sample mean for the Total Responsibility score and overall readiness item will be calculated (range 1-4)
Time Frame: Baseline, Time 2 (about 2 months since baseline), Time 3 (about 5 months since baseline), Time 4 (about 12 months since baseline).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline RTQ Total | 2.73 (0.63) | 2.83 (0.54)
  Time 2 RTQ Total | 3.1 (0.67) | 3.08 (0.49)
  Time 3 RTQ Total | 3.02 (0.72) | 3.07 (0.64)
  Time 4 RTQ Total | 3.16 (0.64) | 3.23 (0.63)
  Baseline RTQ Overall readiness | 2.36 (0.76) | 2.8 (0.96)
  Time 2 RTQ Overall readiness | 2.64 (0.85) | 2.76 (0.97)
  Time 3 RTQ Overall readiness | 2.86 (0.77) | 2.8 (0.91)
  Time 4 RTQ Overall readiness | 3.14 (0.79) | 3.04 (0.95)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.59, Mixed Models Analysis; A linear mixed model for repeated measures was used. The group x time interaction evaluated the effect of the intervention over time
Statistical Analysis 2: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.003, Mixed Models Analysis; A linear mixed model for repeat measures was used. The group x time interaction evaluated the effect of the intervention over time

10. Secondary Outcome: Knowledge (Young Adult Survivors)
Description: The knowledge subscale from the Transition Readiness Inventory (TRI) measures knowledge of survivorship care using a 5-point scale, with higher scores indicating greater knowledge. A mean score will be calculated (range 1-5).
Time Frame: Baseline, Time 2 (about 2 months since baseline), Time 3 (about 5 months since baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.44 (0.71) | 3.9 (0.76)
  Time 2 | 4.1 (0.67) | 4.13 (0.68)
  Time 3 | 4.4 (0.7) | 4.45 (0.77)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.03, Mixed Models Analysis; [statistical method as in outcome 9, analysis 2]

11. Secondary Outcome: Self-Management Skills/Self-Efficacy (Young Adult Survivors)
Description: The Skills/Self-Efficacy sub-scale from the Transition Readiness Inventory (TRI) measures self-management skills and self-efficacy for survivorship care using a 5-point scale, with higher scores indicating greater skills/efficacy. A mean score will be calculated (range 1-5).
Time Frame: Baseline, Time 2 (about 2 months since baseline), Time 3 (about 5 months since baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.4 (0.68) | 3.81 (0.71)
  Time 2 | 3.72 (0.78) | 3.92 (0.66)
  Time 3 | 3.84 (0.76) | 4.00 (0.77)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.07, Mixed Models Analysis; [statistical method as in outcome 9, analysis 2]

12. Secondary Outcome: Self-Management Goals (Young Adult Survivors)
Description: The Goals subscale from the Transition Readiness Inventory (TRI) measures self-management goals for survivorship care using a 5-point scale, with higher scores indicating greater goals. A mean score will be calculated (range 1-5).
Time Frame: Baseline, Time 2 (about 2 months since baseline), Time 3 (about 5 months since baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.44 (0.91) | 3.99 (1)
  Time 2 | 4.10 (0.71) | 4.30 (0.72)
  Time 3 | 4.06 (0.67) | 4.30 (0.89)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.2, Mixed Models Analysis; [statistical method as in outcome 9, analysis 2]

13. Secondary Outcome: Self-Management Beliefs (Young Adult Survivors)
Description: The Beliefs/Expectations sub-scale from the Transition Readiness Inventory (TRI) measures self-management beliefs for survivorship care using a 5-point scale, with higher scores indicating more positive beliefs. A mean score will be calculated (range 1-5).
Time Frame: Baseline, Time 2 (about 2 months since baseline), Time 3 (about 5 months since baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.59 (0.58) | 3.95 (0.64)
  Time 2 | 4.14 (0.45) | 4.06 (0.66)
  Time 3 | 4.21 (0.55) | 4.13 (0.67)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.006, Mixed Models Analysis; [statistical method as in outcome 9, analysis 2]

14. Secondary Outcome: Self-efficacy for Communicating With Physician (Young Adult Survivors): Scale
Description: This single item measures confidence in communicating with a physician about health concerns using a 10-point scale, with higher scores indicating greater confidence. Range is from 1-10.
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 7.89 (1.76) | 8.28 (2.16)
  Time 2 | 8.74 (1.2) | 8.82 (1.77)
  Time 3 | 8.56 (1.35) | 8.92 (1.88)
  Time 4 | 8.67 (1.19) | 9.0 (1.27)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.86, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]

15. Secondary Outcome: Self-efficacy for Communicating With Family About Healthcare (Young Adult Survivors): Scale
Description: This scale measures confidence in communicating with family about healthcare concerns using a 5-point scale, with higher scores indicating greater confidence. A mean score is calculated (range from 1-5).
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.49 (1.04) | 3.96 (1.03)
  Time 2 | 4.08 (1.03) | 4.09 (1.15)
  Time 3 | 3.91 (1.23) | 4.36 (1.03)
  Time 4 | 4.29 (0.89) | 4.19 (0.92)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.14, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]

16. Secondary Outcome: Self-efficacy for Managing Late Effects (Young Adult Survivors): Scale
Description: This scale consists of three items measuring confidence in managing late effects using a 5-point scale, with higher scores indicating higher confidence. A mean score is calculated (range 1-5).
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 2.39 (1) | 3.05 (1.35)
  Time 2 | 3.43 (1.12) | 3.63 (1.18)
  Time 3 | 3.67 (0.97) | 3.65 (1.14)
  Time 4 | 3.7 (0.87) | 3.54 (1.27)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.02, Mixed Models Analysis; A linear mixed model for repeated measures was used. The group x time interaction evaluated the effect of intervention over time

17. Secondary Outcome: Self-efficacy for Survivorship Care Planning (Young Adult Survivors): Scale
Description: This scale consists of three items measuring confidence in survivorship care planning using a 5-point scale, with higher scores indicating higher confidence. A mean score is calculated (range 1-5).
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 2.83 (1.21) | 3.25 (1.53)
  Time 2 | 3.89 (0.89) | 3.65 (1.28)
  Time 3 | 3.92 (1.15) | 3.96 (1.33)
  Time 4 | 4.1 (0.84) | 3.96 (1.18)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.29, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]

18. Secondary Outcome: Health Insurance Self-efficacy (Young Adult Survivors): Scale
Description: This scale consists of seven items measuring confidence in managing health insurance using a 5-point scale, with higher scores indicating higher confidence. A mean score is calculated (range 1-5).
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 2.2 (0.88) | 2.8 (1.22)
  Time 2 | 3.06 (1.25) | 3.01 (1.18)
  Time 3 | 3.45 (1.19) | 3.55 (1.13)
  Time 4 | 3.36 (0.84) | 3.43 (1.17)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.13, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]

19. Secondary Outcome: Survivorship Care Attitudes (Young Adult Survivors)
Description: This scale consists of four items measuring attitudes toward survivorship care using a 5-point scale, with higher scores indicating more positive attitudes. A mean score is calculated (range 1-5).
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 4.07 (0.62) | 3.99 (0.76)
  Time 2 | 4.35 (0.66) | 4.03 (0.93)
  Time 3 | 4.43 (0.57) | 4.25 (0.73)
  Time 4 | 4.54 (0.41) | 4.2 (0.74)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.14, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]

20. Secondary Outcome: Self-efficacy for Managing Emotions (Young Adult Survivors): Scale
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions - Managing Emotions-Short Form is an 8-item measure of confidence in managing emotions. A mean score will be calculated (range 1-5). Higher scores indicate higher confidence in managing emotions.
Time Frame: Baseline, Time 2 (about 2 months since baseline), Time 3 (about 5 months since baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.39 (0.9) | 3.73 (0.87)
  Time 2 | 3.85 (0.94) | 3.73 (0.88)
  Time 3 | 3.97 (0.82) | 3.86 (0.76)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.03, Mixed Models Analysis; [statistical method as in outcome 9, analysis 2]

21. Secondary Outcome: Emotional Support (Young Adult Survivors)
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support-Short Form is a 4-item measure of perceived emotional support. A mean score will be calculated (range 1-5), with higher scores indicative of having better perceived emotional support.
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 4.18 (0.98) | 4.47 (0.77)
  Time 2 | 4.36 (1.04) | 4.5 (0.76)
  Time 3 | 4.3 (1.09) | 4.5 (0.68)
  Time 4 | 4.42 (0.75) | 4.57 (0.63)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.66, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]

22. Secondary Outcome: Informational Support (Young Adult Survivors)
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Informational Support-Short Form is a 4-item measure of perceived availability of helpful information or advice. A mean score will be calculated (range 1-5), with higher scores indicating higher perceived informational support.
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 3.99 (0.94) | 4.35 (0.68)
  Time 2 | 4.41 (0.97) | 4.4 (0.74)
  Time 3 | 4.23 (1.05) | 4.43 (0.71)
  Time 4 | 4.31 (0.71) | 4.29 (0.87)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority; p = 0.15, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]

23. Other Pre Specified Outcome: Healthcare Utilization (Young Adult Survivors)
Description: As an exploratory outcome, participants will report on receipt of the following healthcare (if applicable): Survivorship Care Plan, annual survivorship visit, echocardiogram within last 5 years, mammogram ever (females only), skin cancer screening ever, primary care visit in last 2 years, dental visit in the last year, annual flu vaccine up-to-date, and human papillomavirus (HPV) vaccine ever. Each item will be treated individually. The number of survivors reporting receipt of each healthcare service will be counted. "Yes" indicates receipt within time frame indicated for the outcome; "No" indicates either not received or not due per self-report.
Time Frame: Baseline, Time 3 (about 5 months since baseline), Time 4 (about 12 months since baseline).
Population: Mammogram measure was only administered to females so the sample size for those analyses represent the number of females in each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 25 | 25
Participants
  Survivorship Care Plan-Baseline : yes | 9 | 10
  Survivorship Care Plan-Time 3 : yes | 18 | 15
  Survivorship Care Plan-Time 4 : yes | 18 | 11
  Annual survivorship visit-Baseline: yes | 20 | 16
  Annual survivorship visit-Time 3: yes | 6 | 1
  Annual survivorship visit-Time 4: yes | 15 | 9
  Echocardiogram-Baseline: yes | 19 | 15
  Echocardiogram-Time 3: yes | 19 | 16
  Echocardiogram-Time 4: yes | 18 | 13
  Mammogram-Baseline: yes: number analyzed (Participants) | 11 | 9
  Mammogram-Baseline: yes | 1 | 1
  Mammogram-Time 3: yes: number analyzed (Participants) | 11 | 9
  Mammogram-Time 3: yes | 1 | 1
  Mammogram-Time 4: yes: number analyzed (Participants) | 11 | 9
  Mammogram-Time 4: yes | 1 | 0
  Skin cancer screening-Baseline: yes | 8 | 5
  Skin cancer screening-Time 3: yes | 6 | 7
  Skin cancer screening-Time 4: yes | 8 | 7
  Primary care visit-Baseline: yes | 21 | 24
  Primary care visit-Time 3: yes | 16 | 22
  Primary care visit-Time 4: yes | 19 | 21
  Dental visit-Baseline: yes | 20 | 21
  Dental visit-Time 3: yes | 20 | 17
  Dental visit-Time 4: yes | 15 | 13
  Annual flu vaccine-Baseline | 14 | 12
  Annual flu vaccine-Time 3 | 18 | 17
  Annual flu vaccine-Time 4 | 15 | 16
  Human papillomavirus (HPV) vaccine-Baseline: yes | 19 | 16
  Human papillomavirus (HPV) vaccine-Time 3: yes | 19 | 16
  Human papillomavirus (HPV) vaccine-Time4: yes | 20 | 17

ADVERSE EVENTS:
Time Frame: For the duration of the study - 1 year.
Arm/Group | Intervention | Usual Care | Mentors
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/10
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT04075734/Prot_SAP_001.pdf
  • Informed Consent Form (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT04075734/ICF_000.pdf